CLINICAL TRIAL: NCT03990584
Title: Effects of Irrigation Activation on Clinical Outcomes of Root Canal Treatment in Posterior Teeth With Chronic Apical Periodontitis
Brief Title: Effects of Irrigation Activation on Clinical Outcomes of Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, seydaersahan, Director, Clinical Research, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E34148
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Periapical Periodontitis; Root Canal Infection
Keywords: Chronic apical periodontitis; irrigation activation methods; periapical index; postoperative pain; treatment outcome
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three irrigation activation methods (Experimental): Manual dynamic irrigation was performed using a well-fitting gutta-percha cone inserted to WL with in-and-out vertical strokes of 5 mm at a rate of approximately 100 strokes per minute in order to hydrodynamically displace the irrigant.
  Passive ultrasonic irrigation was performed using a non-cutting size 25 file attached to a piezoelectric ultrasonic unit.
  Sonic irrigation was performed using an EndoActivator sonic handpiece (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA). A suitable-size activator tip was selected and loosely placed at 2 mm from working length, and the device was operated at 10,000 cycles/min using a pumping action to move the tip to produce vertical strokes of 2-3 mm.
  Interventions: Procedure: three irrigation activation methods
- Conventional needle irrigation (control) (Active Comparator): Conventional needle irrigation was performed with short, in-and-out vertical strokes of 2-3 mm at a rate of approximately 100 strokes per minute.
  Interventions: Procedure: conventional needle irrigation

INTERVENTIONS:
Procedure: three irrigation activation methods — passive ultrasonic irrigation, sonic irrigation, manual dynamic irrigation
  Other Names: passive ultrasonic irrigation (Irrisafe; Satelec Acteon, Mérignac, France), sonic irrigation (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA), manual dynamic irrigation (Kerr Dental, USA)
  Arms: three irrigation activation methods
Procedure: conventional needle irrigation — conventional needle irrigation
  Arms: Conventional needle irrigation (control)

SUMMARY:
This study evaluates postoperative pain and radiographic healing of asymptomatic posterior teeth with chronic apical periodontitis following root-canal treatment performed using different methods of irrigation activation.

DETAILED DESCRIPTION:
Aim: To evaluate postoperative pain and radiographic healing of asymptomatic posterior teeth with chronic apical periodontitis following root-canal treatment performed using different methods of irrigation activation.

Methodology: In this prospective clinical trial, root-canal treatment was performed on 162 posterior teeth with chronic apical periodontitis. After routine canal preparation, patients were assigned to either a control group treated using conventional needle irrigation (CNI) without activation or to one of 3 treatment groups, each of which was treated using a different activation protocol during the final irrigation [manual dynamic irrigation (MDI), passive ultrasonic irrigation (PUI), sonic irrigation (SI)]. All treatment was completed in a single visit. Patients provided self-assessments of the severity of postoperative pain at 24h, 48h and 7 days using a modified 4-step visual analogue scale (VAS). Patients were recalled at 12 months for clinical and radiographic examinations. Periodontal healing was evaluated using a periapical index (PAI), with scores of 1 or 2 considered to represent treatment success and scores of 3, 4, or 5 to represent treatment failure. Data were analyzed using one-way ANOVA and Kruskal-Wallis tests, with differences of P < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* a non-contributory medical history
* must have an asymptomatic, necrotic premolar or molar with periapical lesions of > 2.0 x 2.0 mm around one or both roots
* must be diagnosed as chronic apical periodontitis

Exclusion Criteria:

* Those with clinical symptoms (acute pain)
* have periapical radiolucency of >5 mm
* no previous endodontic treatment
* no severe periodontal disease in the related tooth
* non-restorable tooth
* use of any analgesics within the previous 3 days or antibiotics within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
change from baseline postoperative pain at 1 week | 24 hours, 48 hours and 1 week postoperatively
  Pain was measured using a modified visual analogue scale (VAS) with 4 levels, as follows: 1, no pain; 2, slight pain (mild discomfort, no treatment needed); 3, moderate pain (pain required analgesics for relief); 4, severe pain (pain and/or swelling not relieved by simple analgesics and required unscheduled visit). Patients were provided forms and asked to record preoperative pain as well as pain at 24 hours, 48 hours and 1 week postoperatively, and to note down the number of analgesics taken. Patients returned their completed forms at their 1-week follow-up visits.
change from baseline periapical index at 1 year | Clinical and radiographic examinations were performed on the 1 day of treatment,1 day after treatment and 1 year after treatment.
  Periapical tissue was evaluated using a 5-point periapical index (PAI) (Ørstavik et al. 1986) and scored as follows: 1: Normal periapical structures; 2: Small changes in bone structures; 3: Changes in bone structure with some mineral loss; 4: Periodontitis with well-defined radiolucent area; 5: Severe periodontitis with exacerbating features. If scores varied among roots in the same tooth, the highest score was recorded for that tooth. Similarly, if scores varied between observers for the same tooth, the higher score was recorded.
  Treatment was considered successful if the patient had no discomfort, no percussion/palpation pain, no sinus tract, no mobility or associated soft-tissue swelling, and a PAI score of ≤ 2. Treatment was considered a failure if the patient could not perform normal masticatory functions, experienced discomfort and percussive pain upon examination, and/or had a PAI score of ≥ 3 .

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Ersahan, PhD, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After its publication in a journal, we want to share our data
Supporting Information: Study Protocol, SAP
Time Frame: After its publication in a journal, we want to share our data
Access Criteria: postoperative pain scores periapical and panoramic radiographs and radiographic findings clinical findings

REFERENCES:
- [Background] Andrabi SM, Kumar A, Zia A, Iftekhar H, Alam S, Siddiqui S. Effect of passive ultrasonic irrigation and manual dynamic irrigation on smear layer removal from root canals in a closed apex in vitro model. Journal of Investigative and Clinical Dentistry 5: 188-93, 2014. Akerblom A, Hasselgren G. The prognosis for endodontic treatment of obliterated root canals. Journal of Endodontics 14: 565-7, 1998. Attar S, Bowles WR, Baisden MK, Hodges JS, McClanahan SB. Evaluation of pretreatment analgesia and endodontic treatment for postoperative endodontic pain. Journal of Endodontics 34: 652-5, 2008. Brito PR, Souza LC, Machado de Oliveira JC et al. Comparison of the effectiveness of three irrigation techniques in reducing intracanal Enterococcus faecalis populations: an in vitro study. Journal of Endodontics 35: 1422-7, 2009. Brynolf I (1967) A histological and roentgenological study of the periapical region of human upper incisors. Odontologisk Revy 18, 1-176.1-176. Cameron JA (1988) The effect of ultrasonic endodontics on the temperature of the root canal wall. Journal of Endodontics 14, 554-8. Card SJ, Sigurdsson A, Ørstavik D, Trope M . The effectiveness of increased apical enlargement in reducing intracanal bacteria. Journal of Endodontics 28: 779-83, 2002. de Gregorio C, Estevez R, Cisneros R, Heilborn C, Cohenca N . Effect of EDTA, sonic, and ultrasonic activation on the penetration of sodium hypochlorite into simulated lateral canals: an in vitro study. Journal of Endodontics 35: 891-5, 2009. de Gregorio C, Estevez R, Cisneros R, Paranjpe A, Cohenca N . Efficacy of different irrigation and activation systems on the penetration of sodium hypochlorite into simulated lateral canals and up to working length: an in vitro study. Journal of Endodontics 36: 1216-1221, 2010. Desai P, Himel V .Comparative safety of various intracanal irrigation systems. Journal of Endodontics 35: 545-9, 2009.